CLINICAL TRIAL: NCT01965392
Title: Efficiency of an Educational Program for Informal Caregivers of Hospitalized, Dependent Patients: Cluster Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ESCPD-2010
Record Dates: First submitted 2013-10-07; First posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Dependence, Dementias
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- healtn education (Experimental): one group received an educational program
  Interventions: Other: Health education intervention

INTERVENTIONS:
Other: Health education intervention — 'Health education intervention'

SUMMARY:
The aim was to assess whether nursing interventions based on Health Educational Programs for primary informal caregivers of dependent patients may improve their quality of life, decreasing emotional burden and increasing caregiving knowledge, in order to better meet patients' basic needs.

ELIGIBILITY:
Inclusion Criteria:

* Primary informal caregivers of dependent patients, admitted in 30 hospital units, with expected hospital stays of at least one week. A dependent patient is understood to require the aid of someone else in order to carry out basic daily activities.

Exclusion Criteria:

* caregivers with cognitive deficits that could be an obstacle for adequate verbal understanding, illiteracy, persons taking part in other clinical trials or who had taken part in similar workshops in the previous two years, as well as health professionals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
life quality | Data were evaluated with an average one month after discharge, a maximum in September 2009

SECONDARY OUTCOMES:
Caregiver´s burden | Data were evaluated with an average one month after discharge, a maximum in September 2009